CLINICAL TRIAL: NCT06089031
Title: A Prospective Multicenter Registry on Coronary Function Tests, Organized by the Belgian Working Group on Coronary Microcirculation/Belgian Microcirculation Registry.
Brief Title: Belgian Registry on Coronary Function Testing
Acronym: BELmicro
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-0522
Record Dates: First submitted 2023-10-12; First posted 2023-10-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Coronary Microvascular Dysfunction; Coronary Artery Vasospasm
MeSH Terms: conditions — Coronary Vasospasm

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BELmicro: No intervention foreseen.
  Interventions: Diagnostic Test: Coronary Function Test

INTERVENTIONS:
Diagnostic Test: Coronary Function Test — Coronary function test may comprise of bolus thermodilution measurements of coronary microvascular function and/or acetylcholine-derived coronary vasoreactivity tests.

SUMMARY:
The goal of this prospective, multicenter registy is to describe the 'real-world' use of coronary function tests, which may consist of bolus thermodilution measurements of coronary microvascular function and/or invasive vasoreactivity tests with acetylcholine, in the current Belgian routine practice. The main questions it aims to answer are:

* how frequent are coronary function tests performed
* what is the indication for coronary function tests
* what is the frequency of coronary microvascular dysfunction
* what is the frequency of coronary artery vasospasm

From each participant, data will be collected from their medical files concerning cardiovascular risk factors, relevant past medical history, non-invasive tests, procedural data, and follow-up data from routine in-patient visits. Their are no specific study visits. Optionally, patients will be asked to fill in questionnaires about anginal symptoms and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled for coronary function test, comprising of intracoronary bolus thermodilution measurements of microvascular function, and/or intracoronary vasoreactivity tests with acetylcholine.
* Subject understands the study requirements and provides written informed consent.

Exclusion Criteria:

* Subject is participating in another investigational clinical trial that may cause non-compliance with the protocol or confound data interpretation.
* Subject intends to participate in another investigational clinical trial that may cause non-compliance with the protocol or confound data interpretation.
* Documented or suspected pregnancy.
* Inability to provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Current registry includes each patient in which coronary function tests are performed. The indication for coronary function tests is left to the descretion of the operator. The study population will be broader than the classic use of coronary function tests for angina and non-obstructive coronary arteries (ANOCA).
Sampling Method: Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2021-10-18 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of coronary microvascular dysfunction and/or coronary artery vasospasm | 5 years
  To measure the frequency of coronary microvascular dysfunciton coronary artery and vasomotor disorders among patients undergoing coronary function tests.

SECONDARY OUTCOMES:
Describe predictors for coronary microvascular dysfunction and/or coronary artery vasospasm | 5 years
  To find predictors for coronary microvascular dysfunction and/or coronary artery vasospasm by means of multivariate regression analysis.
Describe 1- year and 3-year MACE among the different endotypes of coronary microvascular dysfunction with/whithout coronary artery spasm. | 5 years
  To describe the difference in 1-year and 3-year MACE between the different endotypes of coronary microvascular dysfunction obtained.

CONTACTS AND LOCATIONS:
Locations (13):
- Belgium (13):
  - AZ Monica, Deurne, Antwerp
  - AZ Sint-Maarten, Mechelen, Antwerp
  - Jessa Hasselt, Hasselt, Limburg
  - OLV Aalst, Aalst
  - Ziekenhuis aan de Stroom (ZAS), Antwerp
  - University Hospital Antwerp, Antwerp
  - AZ Sint-Jan Brugge, Bruges
  - AZ Jan Yperman, Ieper
  - AZ Groeninge, Kortrijk
  - UZ Leuven, Leuven
  - CHC Montlégia Liège, Liège
  - CHR Citadelle Liège, Liège
  - AZ Delta, Roeselare

IPD SHARING:
Plan to Share IPD: No